CLINICAL TRIAL: NCT00534586
Title: Influence of Anesthetics on Sedation and Antinociception: an Analysis of Auditory Evoked, Visceral Evoked and Heat Evoked Potentials
Brief Title: Anesthetics and Auditory, Visceral, and Heat Evoked Potentials
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 603/01
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2005-12

CONDITIONS: Healthy
Keywords: Pain; SSEP; CHEPS; Propofol; Sevoflurane; S-Ketamine; Remifentanil; Healthy volunteers
MeSH Terms: conditions — Pain | interventions — Propofol; Remifentanil; Esketamine; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): remifentanil
  Interventions: Drug: Remifentanil
- 2 (Active Comparator): propofol
  Interventions: Drug: Propofol
- 3 (Active Comparator): sevoflurane
  Interventions: Drug: Sevoflurane
- 4 (Active Comparator): s-ketamine
  Interventions: Drug: S-Ketamine

INTERVENTIONS:
Drug: Propofol — TCI 0.5 mcg/ml 1.0 mcg/ml
  Arms: 2
Drug: Remifentanil — continuous infusion 0.05 mcg/kg/min 0.15 mcg/kg/min
  Arms: 1
Drug: S-Ketamine — continuous infusion 0.25 mg/kg/h 0.50 mg/kg/h
  Arms: 4
Drug: Sevoflurane — via face mask 0.40 Vol% 0.80 Vol%
  Arms: 3

SUMMARY:
The aim of the present study is to investigate and quantify the influence of commonly used anesthetics on auditory and pain evoked potentials.

DETAILED DESCRIPTION:
During surgery patients are exposed to different auditory and sensory stimuli. In this study we investigate the influence of different anesthetics to alertness and nociception. In addition to auditory stimuli (AEP as a measure of sedation), Contact Heat Evoked Potential Stimuli (CHEPS), and esophageal evoked potentials from the lower 1/3 of the esophagus are measured to quantify the effects of anesthetics. 60 Volunteers are enrolled into this study. For each drug, three different levels are measured:

* level 1 no medication
* level 2 low dose of medication
* level 3 light sedation dose (volunteer responds to command)

Four drugs are measured in the study:

propofol, sevoflurane, S-ketamine and remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1-2

Exclusion Criteria:

* drugs that effect the central nervous system
* neurological or psychiatric diseases
* contraindications against propofol, sevoflurane, S-ketamine or remifentanil
* any damages or loss of hearing
* heartburn or any stomach diseases

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-12; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
influence of different drugs on evoked responses | 2 hours

SECONDARY OUTCOMES:
discrimination of antinociceptive, visceral-perceptive and sedative effects of anesthetics | 2 hours
quantification of anesthetic components of propofol, sevoflurane, S-ketamine and remifentanil | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Kochs, MD, Study Chair — Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- Technische Universität München, Klinikum rechts der Isar, Department of Anesthesiology, Munich, Bavaria, Germany